CLINICAL TRIAL: NCT05367050
Title: Impact of Daily, Digital and Behavioral Tele-health Tapering Program for Perioperative Surgical Patients Exposed to Opioids.
Brief Title: Impact of a Behavioral Tele-health Program on the Quality of Recovery for Patients Undergoing Total Joint Replacement Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lucid Lane, Inc (Industry)
Collaborators: Stanford University (Other); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 56984
Record Dates: First submitted 2022-04-22; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Opioid Dependence; Opioid Use; Pain, Joint
MeSH Terms: conditions — Opioid-Related Disorders; Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Patients participate in the Lucid Lane therapy program including working with a mental health pain coach for up to 4 weeks before surgery and 4 weeks after surgery.
  All patients receive therapy provided by Lucid Lane, for 4 weeks after surgery
  Interventions: Behavioral: Lucid Lane Therapy Program
- Control (Active Comparator): Patients will participate in a a surgery preparedness course provided by the VA before surgery (Standard of Care) and Lucid Lane therapy after surgery
  All patients receive therapy provided by Lucid Lane, for 4 weeks after surgery
  Interventions: Behavioral: Lucid Lane Therapy Program; Behavioral: Surgical Preparedness Course

INTERVENTIONS:
Behavioral: Lucid Lane Therapy Program — This intervention is designed to aid participants with pre-surgery anxiety management and surgery prep and pain management post-surgery. Participants will be assigned a Lucid Lane pain coach who will utilize mindfulness, cognitive behavioral therapy, group therapy, and mind-body therapies, to accomplish those goals.
Behavioral: Surgical Preparedness Course — This intervention is designed to help the participant prepare for their upcoming surgery. Classes will include discussions around managing chronic pain before surgery, building mental resilience, dealing with the uncertainty of a new diagnosis or treatment plan, questions to ask their anesthesiologist before and on the day of surgery, what to expect during their potential stay at the hospital, and how to optimize their recovery after surgery. Sessions will often include expert doctors who focus on surgery and medical management around it.
  Arms: Control

SUMMARY:
The quality of recovery after surgery is multi-factorial and includes both physical and mental factors. Persistent pain after surgery is a common problem after major surgery and can result in persistent opioid use. The investigators will be evaluating if the addition of a pain coach/councilor before and after surgery, through a tele health platform (LucidLane) can improve participant's recovery from major joint surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 21-90 years old
* Patient is opioid naive i.e hasn't used opioid medication for 30 days prior to surgery
* Patient willing to use Lucid Lane program to provide behavioral health support for up to 4 weeks before surgery and 4 weeks after surgery.
* Patient is willing to discuss Lucid Lane progress with Palo Alto VA's medical team and prescribing clinicians.
* Patient is willing to sign a Lucid Lane Client Agreement.
* Patient is willing to sign an informed consent form

Exclusion Criteria:

* Serious mental illnesses including schizophrenia-spectrum disorders, severe bipolar disorder, and severe major depression.
* Active suicidal ideations
* Patient is on methadone or buprenorphine for treatment of opioid use disorder(i.e. for treatment of addiction, and not for treatment of pain)
* Patient unwilling to use or not possessing access to a device that allows for video visits(e.g. a smart phone, tablet, or computer)
* Patients who are in palliative care
* Unable to use English to participate in the consent process, the intervention or study assessments.
* Unable to provide informed consent to participate

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) or Hip Injury and Osteoarthritis Outcome Score (HOOS) and | Up to 4 months
  The KOOS and HOOS are questionnaires designed to assess short and long-term patient-relevant outcomes following knee/hip injury. They are self-administered and assess five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee/hip-related quality of life. The scores are normalized on a scale of 0 to 100, where 0 indicates severe problems and 100 indicates no problems.
Change in Pain Catastrophizing scale | Up to 4 months
  The Pain catastrophizing scale (PCS) is a self administered, 13-item questionnaire, used to assess a patient's tendency to magnify the threat value of a pain stimulus. It assess rumination, magnification and helplessness. Responses are recorded on a scale of 0-4, where 0 represents absence of the thought and 4 represents the presence of the thought all the time. The scale has a min score of 0 and a max score of 52. A higher score indicates more pain catastrophizing .
Change in Depression Scores | Up to 4 months
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self administered questionnaire used to screen and monitor the severity of depressive symptoms. It inquires about depressive features, that align with the diagnostic and statistical manual of mental disorders, over the course of 2 weeks. Responses are recorded on a scale of 0-3, where 0 represents absence of the symptom and 3 represents its presence nearly every day.
Change in Anxiety Scores | Up to 4 months
  The General Anxiety Disorder-7 (GAD-7) is a self administered, 7-item questionnaire used to measure general anxiety disorder and its severity. Responses are recorded on a scale of 0-3, where 0 represents an absence of the symptom and 3 represents presence nearly every day.

SECONDARY OUTCOMES:
Percent tapered off opioid (50% MME) | 4 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto Division - VA Palo Alto Health Care System, Palo Alto, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT05367050/ICF_000.pdf